CLINICAL TRIAL: NCT02201342
Title: A Phase I/II Dose Escalation Trial of Udenafil in Adolescents With Single Ventricle Physiology After Fontan Palliation
Brief Title: Pharmacokinetic/Pharmacodynamic Study of Udenafil in Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mezzion Pharma Co. Ltd (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pediatric Heart Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHN-Udenafil-01; U01HL068270 (NIH)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Single Ventricle Heart Disease After Fontan Surgery
Keywords: Fontan; Pharmacokinetics; Pharmacodynamics; Exercise capacity; Maximal Oxygen Consumption; Vascular function; EndoPAT; Myocardial performance
MeSH Terms: interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Udenafil 37.5 mg QD (Experimental): Udenafil 37.5 mg tablet once daily for 5 days
  Interventions: Drug: Udenafil
- Udenafil 37.5 mg BID (Experimental): Udenafil 37.5 mg tablet twice daily for 5 days
  Interventions: Drug: Udenafil
- Udenafil 87.5 mg QD (Experimental): Udenafil 87.5 mg tablet once daily for 5 days
  Interventions: Drug: Udenafil
- Udenafil 87.5 mg BID (Experimental): Udenafil 87.5 mg tablet twice daily for 5 days
  Interventions: Drug: Udenafil
- Udenafil 125 mg QD (Experimental): Udenafil 125 mg tablet once daily for 5 days
  Interventions: Drug: Udenafil
- No Drug (No Intervention): Cohort undergoing exercise test only

INTERVENTIONS:
Drug: Udenafil — Drug
  Arms: Udenafil 125 mg QD; Udenafil 37.5 mg BID; Udenafil 37.5 mg QD; Udenafil 87.5 mg BID; Udenafil 87.5 mg QD

SUMMARY:
To determine the pharmacokinetic profile and safety of udenafil in adolescents with Fontan physiology and to assess the short-term pharmacodynamic effect of udenafil on pharmacodynamic measures of exercise capacity, ventricular performance, and vascular function.

DETAILED DESCRIPTION:
A dose escalation trial to determine the pharmacokinetics, safety and tolerance of udenafil in male and female adolescent subjects with single ventricle physiology that that have undergone the Fontan surgical procedure. Pharmacodynamic data will also be collected to evaluate the effect of udenafil on acute exercise performance, peripheral vascular function and indices of myocardial performance. Five udenafil cohorts will be evaluated in additional to one drug free cohort

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with Fontan physiology who are 14-18 years of age.
2. Willingness to return to center to complete blood draws and exercise tests as described in the study protocol.
3. Patients must agree to abstain from alcohol, caffeinated beverages, and grapefruit juice for the duration of the trial.
4. Informed assent from subject informed consent from parent/legal guardian as appropriate.

Exclusion Criteria:

1. Non-cardiac medical, psychiatric, and/or social disorder that would prevent successful completion of planned study testing or would invalidate its results.
2. Height <132 cm (minimum height requirement for exercise stress testing).
3. Known Fontan baffle obstruction, branch pulmonary artery stenosis, or pulmonary vein stenosis resulting in a mean gradient of >4 mmHg between the regions proximal and distal to the obstruction.
4. Single lung physiology.
5. Severe ventricular dysfunction or valvular regurgitation (systemic atrioventricular or semilunar valve) determined from review of the echocardiogram performed in closest proximity to study enrollment.
6. Significant renal (serum creatinine > 2.0), hepatic (serum aspartate aminotransferase (AST) and/or alanine aminotransferase ( ALT) > 3 times upper limit of normal), gastrointestinal or biliary disorders that could impair absorption, metabolism or excretion of orally administered medications, based on laboratory assessment at the time of screening visit.
7. Hospitalization for acute decompensated heart failure within the 12 months preceding study enrollment.
8. A diagnosis of active protein losing enteropathy or plastic bronchitis.
9. Active evaluation or listing for heart transplant.
10. History of use of a phosphodiesterase type 5 inhibitor within three months of study enrollment.
11. Concurrent illness that, in the opinion of the investigator, precludes participation.
12. Current therapy with alpha-blockers or nitrates.
13. Pregnancy at the time of enrollment.
14. Latex allergy

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Goldberg, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (5):
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Michigan Congenital Heart Center, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Medical Center, Salt Lake City, Utah
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Udenafil 125 mg mg QD: Udenafil 125 mg tablet once daily for 5 days
- No Drug: Only exercise testing
Period: Overall Study
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg mg QD | No Drug
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.0) | 16.2 (0.8) | 15.0 (0.9) | 15.5 (1.8) | 16.5 (1.5) | 16.2 (1.2) | 15.8 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 3 | 2 | 2 | 15
  Male | 4 | 3 | 3 | 3 | 4 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 5 | 5 | 6 | 6 | 6 | 6 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 0 | 0 | 3
  White | 3 | 4 | 6 | 6 | 4 | 5 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 0 | 0 | 3 | 4 | 7
  United States | 6 | 6 | 6 | 6 | 3 | 2 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events Possibly or Probably Related to Udenafil
Description: Number of subjects experiencing serious adverse events possibly or probably related to udenafil at doses of 37.5 mg daily, 37.5 mg twice daily, 87.5 mg daily, 87.5 mg twice daily, and 125 mg daily given over a five-day period.
Time Frame: 5 days
Measure: Number; unit: participants
Groups:
- No Drug: Exercise only
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Udenafil: Cmax
Description: Evaluate the pharmacokinetic (PK) profile of udenafil, by weight, age, and gender in adolescents with Fontan physiology at multiple dosing levels.
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
ng/ml | 94.8 (46.2) | 152 (46.1) | 277 (107) | 506 (188) | 438 (173) |

3. Secondary Outcome: Evaluate the Effect of Udenafil on Pharmacodynamic (PD) Outcomes: Exercise Capacity
Description: Evaluate the effect of udenafil on pharmacodynamic (PD) outcomes including: exercise capacity, vascular function, and echocardiographic measures of myocardial performance (MPI). The outcome measures (OM) are a difference between baseline (BL) and follow-up (FU) [OM = FU-BL].
Time Frame: Day 1 (baseline) and Day 5 (follow-up)
Population: n= 4 to 5 for some measures
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ml/kg/min
  Max VO2 at max exercise effort: number analyzed (Participants) | 5 | 6 | 6 | 5 | 5 | 5
  Max VO2 at max exercise effort | -0.8 (1.7) | -1.6 (5.1) | -1.4 (2.5) | 0.2 (5.0) | 0.9 (2.6) | -0.3 (1.8)
  VO2 at anaerobic threshold: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
  VO2 at anaerobic threshold | -0.5 (4.1) | 0.1 (1.0) | -1.1 (1.9) | -1.7 (2.1) | 1.2 (1.9) | 0.1 (3.8)

4. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Metabolite DA-8164: Cmax
Description: Evaluate the pharmacokinetic (PK) profile of metabolite DA-8164, by weight, age, and gender in adolescents with Fontan physiology at multiple dosing levels.
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
ng/ml | 61.3 (28.4) | 159 (82.0) | 227 (149) | 293 (101) | 256 (32.5) |

5. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Udenafil: Tmax
Description: as for outcome 2
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
hr | 2.25 (0.880) | 1.50 (0.837) | 2.11 (0.735) | 1.25 (0.274) | 1.58 (0.665) |

6. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Udenafil: T-1/2
Description: as for outcome 2
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
hr | 12.9 (3.12) | 13.3 (1.48) | 12.6 (0.897) | 10.4 (1.19) | 11.1 (2.80) |

7. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Udenafil: AUC (0-tau)
Description: as for outcome 2
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
hr*ng/ml | 834 (403) | 1050 (387) | 2200 (459) | 3350 (796) | 3420 (1800) |

8. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Udenafil: CLSS/F
Description: as for outcome 2
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: l/hr
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
l/hr | 53.3 (21.3) | 39.9 (14.2) | 41.1 (7.76) | 27.2 (5.39) | 43.3 (16.8) |

9. Secondary Outcome: Evaluate the Effect of Udenafil on Pharmacodynamic (PD) Outcomes: Vascular Function [Change in Natural Log Transformed Reactive Hyperemia Index (RHI)]
Description: Evaluate the effect of udenafil on pharmacodynamic (PD) outcomes including: exercise capacity, vascular function, and echocardiographic measures of myocardial performance (MPI). The outcome measures (OM) are a difference between baseline (BL) and follow-up (FU, Day-5) [OM = FU-BL]. Endothelial pulse amplitude tonometry (Endo-PAT) is a technique for the non-invasive assessment of peripheral vascular function. In adults, Endo-PAT has been demonstrated to identify those with coronary artery dysfunction and to correlate with brachial artery reactivity testing. Endo-PAT use in children has been more limited, but has shown excellent reproducibility. Reactive hyperemia index (RHI), a measure of the hyperemic response adjusted for baseline blood flow, is a measure of vascular function. A higher value denotes better, or more healthy, vascular (endothelial) function. The data represents a change in the index value so there is no minimum or maximum value that can be represented on a scale.
Time Frame: Day 1 (baseline) and Day 5 (follow-up)
Population: n= 4 to 5 for some measures
Measure: Mean (Standard Deviation); unit: Change in natural log Transformed RHI
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 6 | 0
Change in natural log Transformed RHI | 0.3 (0.47) | -0.07 (0.17) | 0.07 (0.22) | -0.03 (0.20) | -0.10 (0.38) |

10. Secondary Outcome: Absolute Change in Blood Pool Myocardial Performance Index (MPI)
Description: The outcome measures (OM) are a difference between baseline (BL) and follow-up (FU, Day-5). Change in the MPI from baseline to Day 5 is determined by velocities from blood pool Doppler of the inflow and outflow tract of the dominant ventricle. The measure is the ratio of the sum of isovolumetric contraction time and isovolumetric relaxation time, divided by ventricular ejection time. A lower value is consistent with a more efficient ventricle (better function). A value of zero indicates that there is no isovolumetric contraction or relaxation and, while physiologically implausible, would be consistent with a perfectly efficient ventricle. In general, a decrease in the MPI corresponds to more efficient (better) ventricular function, while an increase in MPI corresponds to less efficient (worse) ventricular function. The data represents a change in the index value so there is no minimum or maximum value that can be represented on a scale.
Time Frame: Day 1 (baseline) and Day 5 (follow-up)
Population: n= 4 to 5 for some measures
Measure: Mean (Standard Deviation); unit: Change in blood pool MPI
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 5 | 0
Change in blood pool MPI | -0.052 (0.166) | -0.003 (0.102) | -0.076 (0.144) | -0.118 (0.090) | -0.054 (0.180) |

11. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Metabolite DA-8164: Tmax
Description: as for outcome 4
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0
hr | 3.08 (1.56) | 2.09 (1.62) | 3.19 (0.949) | 2.58 (0.917) | 3.84 (1.33) |

12. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Metabolite DA-8164: T-1/2
Description: as for outcome 4
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 4 | 0
hr | 15.9 (4.90) | 14.4 (2.31) | 15.3 (2.73) | 12.6 (2.25) | 14.7 (2.30) |

13. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of Metabolite DA-8164: AUC(0-tau)
Description: as for outcome 4
Time Frame: Day 5, zero to 48 hours after the last dose
Population: The No Drug Group is not eligible for PK analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 0
hr*ng/ml | 881 (375) | 1290 (710) | 2910 (1880) | 2410 (568) | 3470 (471) |

ADVERSE EVENTS:
Arm/Group | Udenafil 37.5 mg QD | Udenafil 37.5 mg BID | Udenafil 87.5 mg QD | Udenafil 87.5 mg BID | Udenafil 125 mg QD | No Drug
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 6/6 | 5/6 | 6/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Udenafil 37.5 mg QD (N=6) | Udenafil 37.5 mg BID (N=6) | Udenafil 87.5 mg QD (N=6) | Udenafil 87.5 mg BID (N=6) | Udenafil 125 mg QD (N=6) | No Drug (N=6)
Altered mental status/mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related to the study drug, per PI.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Udenafil 37.5 mg QD (N=6) | Udenafil 37.5 mg BID (N=6) | Udenafil 87.5 mg QD (N=6) | Udenafil 87.5 mg BID (N=6) | Udenafil 125 mg QD (N=6) | No Drug (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flushing (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 4 (4) | 2 (7) | 1 (1) | 0 (0)
Headache (General disorders) | 3 (9) | 4 (6) | 4 (9) | 4 (12) | 5 (14) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (6) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other